CLINICAL TRIAL: NCT04873609
Title: Targeted Electronic Patient Portal Messaging Increases Hepatitis C Virus Screening in Primary Care: a Randomized Study
Brief Title: Electronic Record Assimilation and Subsequent Eradication of Hepatitis C
Acronym: ERASE-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Aparna Goel, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: eP46287
Record Dates: First submitted 2021-04-22; First posted 2021-05-05 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Hepatitis C; Liver Diseases
Keywords: Hepatitis C screening; Population Health
MeSH Terms: conditions — Hepatitis C; Liver Diseases | interventions — Community-Institutional Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No primary care provider (PCP) appointment, No patient outreach (No Intervention): 400 patients that did not have an upcoming PCP appointment in 6 months were randomly assigned to control group and did not receive a patient portal message with order for HCV antibody screening
- No PCP appointment, Patient outreach (Active Comparator): 400 patients that did not have an upcoming PCP appointment in 6 months were randomly assigned to receive a patient portal message with order for HCV antibody screening
  Interventions: Behavioral: Patient portal message
- PCP appointment, No patient outreach (No Intervention): 400 patients that had an upcoming PCP appointment in 6 months were randomly assigned to control group and did not receive a patient portal message with order for HCV antibody screening
- PCP appointment, Patient outreach (Active Comparator): 400 patients that had an upcoming PCP appointment in 6 months were randomly assigned to receive a patient portal message with order for HCV antibody screening
  Interventions: Behavioral: Patient portal message

INTERVENTIONS:
Behavioral: Patient portal message — Direct-to-patient message via the electronic patient portal (MyHealth) with HCV antibody lab order directed to their preferred laboratory
  Other Names: outreach
  Arms: No PCP appointment, Patient outreach; PCP appointment, Patient outreach

SUMMARY:
Given the disproportionately high risk of chronic hepatitis C virus (HCV) infection in the baby boomer cohort, population-based screening has been demonstrated cost effective. Compared to point-of-care testing, however, bulk health messages with coupled lab requisitions delivered directly to patients meeting screening criteria via patient portals could improve HCV screening at minimal cost.

DETAILED DESCRIPTION:
The Centers for Disease Control and Prevention (CDC) and the United States Preventative Services Taskforce (USPSTF) recommend a one-time hepatitis C infection (HCV) screen in individuals born 1945-65 (baby boomer birth cohort) and in others with risk factors for infection. National adherence to this Grade B recommendation-carrying the same strength of evidence as mammography, and screening for depression, alcohol abuse, and type 2 diabetes-is estimated to be 13.8%. Efforts to increase screening and linkage to HCV care, and also to understand barriers to screening and linkage are therefore warranted.

One such intervention, direct-to-patient messages via electronic medical record (EMR), has been demonstrated to improve adherence in influenza and pneumococcal vaccination, colon cancer screening, immunosuppression after transplantation, among others, but has not been studied as a strategy to improve HCV screening rates within health systems.

Our institution, Stanford Health Care, comprises 86 distinct clinical sites with approximately 1.25 million outpatient visits per year. All clinical sites are linked with an EMR (Epic Systems Corp.) and patients are encouraged to opt-in to receive and send health-related messages through a secure internet and smartphone portal, MyHealth. Approximately 60% of patients at our institution are enrolled in MyHealth.

MyHealth additionally allows bulk-messaging of patients meeting specific characteristics, e.g. patients due for influenza vaccination. Bulk messages can be coupled with laboratory or radiology requisitions. Messages are delivered through the online portal, text message, e-mail, and/or smartphone application notification, depending on patient preference. Laboratory and radiology results are routed automatically to patients' primary care physicians for review.

The investigators propose to conduct a randomized study comparing the effectiveness of a direct-to-patient electronic health message on HCV screening coupled with a lab requisition, versus HCV screening initiated by primary care clinicians as part of routine clinical care alone.

ELIGIBILITY:
Inclusion Criteria:

* persons born between 1945-1965
* having an activated patient portal to receive secure messages (MyHealth)
* no prior HCV antibody test within our EHR (electronic health record), including externally accessible results

Exclusion Criteria:

* documented HCV viral load in our EHR
* diagnosis of chronic HCV in their problem list

Ages: 54 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Rate of HCV antibody test completion | 6 months
  completion of HCV antibody test

SECONDARY OUTCOMES:
Rate of positive HCV antibody or positive HCV RNA referred for treatment | 8 months
  referral to subspecialty for treatment of chronic HCV infection
Rate of subspecialty visit completion | 3 months
  attended subspecialty visit for treatment
Rate of HCV treatment initiation | 10 months
  chronic HCV treatment started
Rate of sustained virologic response | 10 months
  HCV cured

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Goel, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared.